CLINICAL TRIAL: NCT05901831
Title: A Parallel-group, Randomized, Prospective, Interventional, Double-blind, Multicenter Global Phase 3 Study to Investigate the Efficacy and Safety of Finerenone Versus Placebo, in Addition to Standard of Care, in Participants With Chronic Kidney Disease and Type 1 Diabetes
Brief Title: A Study to Learn How Well the Study Treatment Finerenone Works and How Safe it is in People With Long-term Decrease in the Kidneys' Ability to Work Properly (Chronic Kidney Disease) Together With Type 1 Diabetes
Acronym: FINE-ONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22267; 2022-503024-27-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 1 | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Finerenone arm (Experimental): Participants with eGFR ≥25 to <60 mL/min/1.73 m^2 at Screening visit will take Finerenone Dose A. Participants with eGFR ≥60 mL/min/1.73 m^2 at Screening visit will take Dose B. Up-titration and down-titration of study intervention will be based on local potassium and kidney function (eGFR) values. Treatment duration is 6 months.
  Interventions: Drug: Finerenone
- Placebo arm (Placebo Comparator): Participants will take Finerenone matching placebo for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Finerenone — Dose A, Dose B, oral
  Arms: Finerenone arm
Other: Placebo — Oral
  Arms: Placebo arm

SUMMARY:
Researchers are looking for a better way to treat people with chronic kidney disease (CKD), a progressive decrease in the kidneys' ability to work properly, and type 1 diabetes.

In people with type 1 diabetes, the body does not make enough of a hormone called insulin, resulting in high blood sugar levels that can cause damage to the kidneys. CKD often occurs together with or as a consequence of type 1 diabetes.

The study treatment finerenone works by blocking certain proteins, called mineralocorticoid receptors. An increased stimulation of these proteins is thought to damage the kidneys and the heart. By lowering their stimulation, finerenone reduces the risk of kidney disease progressively getting worse. Finerenone is approved for doctors to prescribe to people with CKD and type 2 diabetes.

In this study, researchers want to learn if finerenone works better than placebo in reducing the participants' kidney disease from getting worse when given in addition to standard of care (SOC) treatment. A placebo looks like a treatment but does not have any medicine in it. SOC is a procedure or treatment that medical experts consider most appropriate for a condition or disease. To find out how well finerenone works, the level of a protein (albumin) in the urine will be measured.

Researchers also want to know how safe finerenone is. To do this, the researchers will collect the number of participants with:

* medical problems (also called treatment-emergent adverse events (TEAEs))
* serious TEAEs. An TEAE is considered 'serious' when it leads to death, puts the participant's life at risk, requires hospitalization, causes disability, causes a baby being born with medical problems, or is medically important
* higher than normal blood levels of potassium (hyperkalaemia). Depending on the treatment group, the participants will either take finerenone or placebo, Importantly, the participants will also continue to take their regular SOC medicines.

The participants will be in the study for up to 7.5 months and will take the study treatments for 6 months. During the study, they will visit the study site at least 6 times.

The study team will:

* collect blood and urine samples
* check the participants' vital signs such as blood pressure and heart rate
* do a physical examination including height and weight
* check the participants' heart health by using an electrocardiogram (ECG)
* do pregnancy tests in women of childbearing potential

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age (or the legal age of consent according to local legislation) at the time of signing the informed consent.
* Participants with Type 1 diabetes (T1D), i.e. T1D continuously treated with insulin, started within one year from diagnosis.

  * If the onset was after age 35, documentation of the presence of one or more of the following:

    * Circulating T1D-associated autoantibodies
    * Hospitalization for diabetic ketoacidosis
    * Plasma C-peptide below the limit of detection with standard assay (with concurrent blood glucose >100 mg/dl).
* HbA1c at Screening <10% (central assessment).

  * Note: One reassessment is allowed for HbA1c during the Screening period in case the first measurement is missing/unreadable/invalid.
* K+ ≤ 4.8 mmol/L at Screening (local assessment)
* Participants with a clinical diagnosis of CKD and fulfilling both the criteria (central assessment):

  * eGFR ≥25 and <90 mL/min/1.73 m^2 using CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) 2009 formula at the Screening visit
  * UACR ≥200 mg/g (22.6 mg/mmol) to <5000 mg/g (565 mg/mmol) at the Screening visit (geometric mean of the 3 measurements)
* Participants on a stable (preferably without any change in the dosage for at least 4 weeks prior to the Screening visit) ACEI (Angiotensin-converting enzyme inhibitor) or ARB (Angiotensin receptor blocker) treatment.

Exclusion Criteria:

* Participant with T2D (Type 2 diabetes).
* Participant with mean BP (Blood pressure) higher than 160/100 mmHg or mean systolic BP lower than 90 mmHg at the Screening visit
* Symptomatic heart failure with reduced ejection fraction with class 1A indication for Mineralocorticoid receptor antagonists (MRAs).
* Participants with current or previous (within 8 weeks prior to the Screening visit) treatment with a SGLT-2/-1 (Sodium-Glucose co-transporter-2/-1) inhibitor or GLP1 (Glucagon-like peptide-1) receptor agonist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Urinary albumin-to-creatinine ratio (UACR) | From baseline up to 6 months
  UACR will be assessed by the Central laboratory.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), Treatment-emergent serious adverse event (TESAEs) | From baseline up to 7 months
Number of participants with Hyperkalaemia | From baseline up to 7 months
  Hyperkalemia will be an adverse events of special interest (AESI).

CONTACTS AND LOCATIONS:
Locations (80):
- United States (28):
  - Southwest Kidney Institute, PLC - Suprise, Surprise, Arizona
  - Stanford Endocrinology Clinic, Stanford, California
  - Touro University California - Metabolic Research Center, Vallejo, California
  - UHealth Diabetes Research Center, Miami, Florida
  - AdventHealth Translational Research Institute, Orlando, Florida
  - Elixia Central Florida, Orlando, Florida
  - Hanson Clinical Research Center, Inc., Port Charlotte, Florida
  - Jedidiah Clinical Research, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Grady Memorial Hospital - Endocrinology, Atlanta, Georgia
  - Northwestern University | Feinberg School of Medicine - Division of Endocrinology, Metabolism and Molecular Medicine, Chicago, Illinois
  - UChicago Medicine Kovler Diabetes Center, Chicago, Illinois
  - Preventive Intervention Center - Endocrinology, Iowa City, Iowa
  - Wichita Nephrology Group Pa, Wichita, Kansas
  - Diabetes & Metabolism Associates, Metairie, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - MU Health Care - University Hospital - Endocrinology, Columbia, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - UNC Endocrinology, Diabetes, and Obesity Clinical Research Unit, Chapel Hill, North Carolina
  - Physicians East, P.A.- W. H. Smith - Endocrinology, Greenville, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - OHSU Physicians Pavillion - Endocrinology, Portland, Oregon
  - UT Health San Antonio - Medical Arts & Research Center - Endocrinology, San Antonio, Texas
  - Consano Clinical Research, LLC., San Antonio, Texas
  - EVMS Strelitz Diabetes Center, Norfolk, Virginia
  - Providence Medical Research Center, Spokane Valley, Washington
- Canada (5):
  - Richmond Road Diagnostic and Treatment Centre - Clinical Trials Unit(RRDTC), Calgary, Alberta
  - Alberta Diabetes Institute - Clinical Research Unit (CRU), Edmonton, Alberta
  - Toronto General Hospital - University Health Network, Renal Physiology laboratory, Toronto, Ontario
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - McGill University Health Centre (MUHC) - Research Institute (RI) - McConnell Centre for Innovative Medicine (CIM), Montreal, Quebec
- China (12):
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The 4th Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Central Hospital of Wuhan, Tongji Medl Collg Huazhong..., Wuhan, Hubei
  - Affiliated Hospital of Jiangsu University, JiangSu, Jiangsu
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Peking University People's Hospital, Beijing
  - Southern Medical University - Nanfang Hospital (Southern Hospital), Guangzhou
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an
  - Nanjing Medical University (NMU) - The Second Affiliated Hospital, Nanjing
  - Shanghai Jiao Tong University (SJTU) - Shanghai General Hospital (Shanghai First People's Hospital) - Northern Location, Shanghai
  - Central Hospital of Minhang District, Shanghai, Shanghai
  - Zhongshan Hospital Fudan University, Qingpu Branch, Shanghai
- Denmark (6):
  - Hospital of South West Jutland | Department of Endocrinology Research, Esbjerg
  - Region Nordjylland | Steno Diabetes Center Nordjylland - Endocrinology Department, Gistrup
  - Steno Diabetes Center Copenhagen | Herlev - Clinical and Translational Research Department, Herlev
  - Region Midtjylland | Regionshospitalet Godstrup - Nephrology Department, Herning
  - Capital Region | Nordsjaellands Hospital - Hillerod - Endocrinology Ambulatory Research Unit, Hillerød
  - Odense University Hospital | Odense - Endocrinology Department, Odense
- Germany (2):
  - InnoDiab Forschung GmbH, Essen, North Rhine-Westphalia
  - Ruhr-Universitaet Bochum - Herz und Diabeteszentrum NRW (Heart and Diabetes Center), Bad Oeynhausen
- Italy (9):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Endocrinologia e prevenzione e cura del diabete, Bologna, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOSD Diabetologia, Rome, Lazio
  - Careggi University Hospital - Diabetologia e Malattie del Metabolismo, Florence, Tuscany
  - ASST Papa Giovanni XXIII | Ospedale di Bergamo - SC Malattie Endocrine-Diabetologia, Bergamo
  - Azienda Sanitaria Locale di Chieri | TO5 - SC Diabetologia Territoriale, Chieri
  - Università degli Studi "G. D'Annunzio" di Chieti - Endocrinologia, Chieti
  - IRCCS Ospedale San Raffaele | Diabetologia Department - Cardio-Metabolic and Clinica Trials Unit, Milan
  - ASST Santi Paolo e Carlo | San Paolo Hospital - Haemostasis and Thrombosis Department, Milan
  - ASST Fatebenefratelli Sacco _Ospedale Sacco - Malattie Endocrine e Diabetologia, Milan
- South Korea (5):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Gerencia de Gestion Integrada A Coruna | Department of Endocrinology and Nutrition, A Coruña, A Coruña
  - Hospital Nisa Sevilla Aljarafe - Endocrinologia, Castilleja de la Cuesta, Sevilla
  - Hospital Clinic de Barcelona | Instituto Clinic de Enfermedades Digestivas y Metabolicas - Endocrinologia y Nutricion, Barcelona
  - Hospital Gregorio Maranon | Endocrinology Department, Madrid
  - Hospital Universitario Puerta De Hierro De Majadahonda - Endocrinologia, Majadahonda
  - Hospital Universitario Virgen De La Victoria - Endocrinologia, Málaga
- United Kingdom (7):
  - North Bristol NHS Trust | Southmead Hospital - Clinical Research Centre, Bristol
  - Cardiff and Vale University Health Board | University Hospital of Wales - Nephrology and Transplant, Cardiff
  - University Hospitals of Derby and Burton NHS Foundation Trust | Royal Derby Hospital - Renal Research, Derby
  - NHS Greater Glasgow and Clyde (NHSGGC) - Glasgow Royal Infirmary (GRI), Glasgow
  - Barts Health NHS Trust - Royal London Hospital - Nephrology, London
  - Manchester University NHS Foundation Trust | Wythenshawe Hospital - Clinical Research Facility, Manchester
  - Walsall Healthcare NHS Trust | Manor Hospital - Nephrology, Walsall

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Kugathasan L, Aronson Y, Sridhar VS, Ni H, Ouimet JP, Limonte CP, Sarma S, Cherney DZI. Advancing kidney protection in type 1 diabetes: insights from emerging therapies in type 2 diabetes and chronic kidney disease. Expert Rev Clin Immunol. 2025 Aug;21(8):1113-1134. doi: 10.1080/1744666X.2025.2537446. Epub 2025 Jul 24. PMID 40693871
- [Derived] Heerspink HJL, Birkenfeld AL, Cherney DZI, Colhoun HM, Ji L, Mathieu C, Groop PH, Pratley RE, Rosas SE, Rossing P, Skyler JS, Tuttle KR, Lawatscheck R, Scott C, Edfors R, Scheerer MF, Kolkhof P, McGill JB. Rationale and design of a randomised phase III registration trial investigating finerenone in participants with type 1 diabetes and chronic kidney disease: The FINE-ONE trial. Diabetes Res Clin Pract. 2023 Oct;204:110908. doi: 10.1016/j.diabres.2023.110908. Epub 2023 Oct 5. PMID 37805000
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22267